CLINICAL TRIAL: NCT03657381
Title: Phase Ⅰ Study to Evaluate the Safety and Tolerability of Using F520 by Advanced Tumor Subjects
Brief Title: Phase Ⅰ Study to Evaluate the Safety and Tolerability of Using F520
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-001
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Advanced Solid Tumor，Recurrent Solid Tumor，Lymphoma，Recurrent Lymphocyte Depleted Classical Hodgkin Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- F520 0.2mg/kg single-dose (Experimental): F520 0.2mg/kg single-dose
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 1.0mg/kg single-dose (Experimental): F520 1.0mg/kg single-dose
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 3.0mg/kg single-dose (Experimental): F520 3.0mg/kg single-dose
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 200mg/times single-dose (Experimental): F520 200mg/times single-dose
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 10mg/kg single-dose (Experimental): F520 10mg/kg single-dose
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 1mg/kg multiple dosing, every 2 weeks (Experimental): F520 1mg/kg every 2 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 3mg/kg multiple dosing, every 2 weeks (Experimental): F520 3mg/kg every 2 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 200mg/times multiple dosing, every 2 weeks (Experimental): F520 200mg/times every 2 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 10mg/kg multiple dosing, every 2 weeks (Experimental): F520 10mg/kg every 2 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 3mg/kg multiple dosing, every 3 weeks (Experimental): F520 3mg/kg every 3 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection
- F520 200mg/times multiple dosing, every 3 weeks (Experimental): F520 200mg/times every 3 weeks
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection

INTERVENTIONS:
Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection — Biological: F520 single-dose:0.2mg/kg, 1.0mg/kg, 3.0mg/kg, 200mg/times, 10mg/kg; multiple dosing: 1mg/kg, 3mg/kg, 200mg/times, 10mg/kg, treat every 2 weeks; multiple dosing: 3mg/kg, 200mg/times, treat every 3 weeks.

SUMMARY:
Recombinant Programmed death-1(PD-1) humanized monoclonal antibody injection (company code: F520) is joint developed by Shandong New Time Pharmaceutical Co., LTD., it is the reorganization of deoxyribonucleic acid (DNA) technology in the Chinese hamster ovary (CHO) cells express system expressed in a immunoglobulin G1 (IgG1) kappa type single resistance to predominate. F520 had the different new amino acid sequence and molecular structure compared with two marketed PD-1 monoclonal antibody injection and got the approval of China Food and Drug Administration (CFDA) for clinical trial.Pharmaceutical research indicated F520 cell strain had security source, production process is stable, quality can control, preparation stability, has good compatibility with packaging materials, it has the condition of industrialization, can prepare investigational medicinal product with safety, effective, and controlled quality for clinical research.Pharmacodynamics study show the targets and mechanisms of F520is clear, tumor suppression effect is obvious.Toxicology studies show this product in high doses with low toxic, and the toxic is reversible, the most common toxicity is specific to the drug action mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-65 years of age;
2. Histologically or cell confirmed advanced, unresectable or metastatic disease tumor and failure to standard therapies or lack of standard therapy(disease progress or failed to tolerate the toxicity, such as chemotherapy, targeted therapy, and other immunotherapies other than PD-1/PD-L1);
3. Agree to provide archived tumor tissue specimens or fresh tissue specimens;
4. ECOG performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks.;
6. At least one measurable and evaluable tumor lesion (in accordance with international working group criteria/RANO/cheson 2007)；
7. Adequate laboratory parameters during the screening period as evidenced by the following（No blood components and cell growth factors are allowed within 28 days prior to screening）:

   routine blood tests: Absolute neutrophil count ≥1.0×109/L ;Platelets ≥100×109/L;Hemoglobin ≥ 9.0 g/dL; Liver function：Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), ALT and AST ≤2.5ULN; for subjects with liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5×ULN, Total bilirubin (TBIL) ≤3×upper limit of normal (ULN); Renal function CCr≤1.5×ULN，Creatinine clearance≥50 mL/min;
8. Thyroid function indicators: thyroid-stimulating hormone (TSH) and free thyroxine (FT3/FT4) are within the normal range;
9. Understand study procedures and contents, and voluntarily sign the written informed consent form.

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: Immune-related neurological diseases, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic lupus erythematosus, connective tissue disease, scleroderma, inflammatory bowel disease including Crowe Enthusiasm and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis or Stevens-Johnson syndrome；
2. Presence of symptomatic central nervous system (CNS) metastases；
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 14 days before entering the group and during the study period;
4. Prior radiotherapy, systemic chemotherapy hormone therapy, surgery or target therapy within 4 weeks or 5 half-lives(whichever is longer) before the study drug administration, or any unresolved AEs > CTC-AE Grade 1;
5. Autologous hematopoietic stem cell transplantation (ASCT) has been completed at least 3 months before receiveing first dose;
6. Known history of hypersensitivity to macromolecular protein preparation or any components of the F520 formulation；
7. Patients receiving any anti-infection vaccine within 4 weeks before enrollment;
8. History or concurrent with other malignant disease, except completely cured basal cell skin cancers and carcinoma in situs of cervix;
9. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) >2 NYHA 2 congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
10. Active infection（needing therapy） or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
11. Patients with active pulmonary tuberculosis; patients who previously had active pulmonary tuberculosis;
12. History of immunodeficiency (HIV) or active hepatitis(Hepatitis B: HBsAg, Anti-HBs, HBeAg, Anti-HBe, Anti-HBc,HBV-DNA; Hepatitis C: Anti-HCV,HCV-RNA)
13. Participation in a clinical study or less than 1 month from the last dose of investigational drug to sign ICF;
14. History of PD-1/PD-L1 or CTLA-4 therapy;
15. Patients with drug abuse history or alcohol addiction history;
16. Patients with current or previous interstitial lung diseases;
17. Female and male who have reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 6 months after receiving the last dose of study treatment.
18. Other factors that may lead to the termination of the participation in the study at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1.5 years

SECONDARY OUTCOMES:
PD-1 receptor occupancy of blood | 3 years
Objective Response Rate (ORR) by irRC/ RECIST 1.1/RANO/cheson2007 | 3 years
Disease Control Rate (DCR) by irRC/ RECIST 1.1/RANO/cheson2007 | 3 years
Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) | 1.5years
Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb | 1.5years
Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb | 1.5years
t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb | 1.5years
Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb | 1.5years
Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb | 1.5years
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5years
Average Plasma Concentration (Cavg) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5years
degree of fluctuation (DF) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5years
Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb | 1.5years

OTHER OUTCOMES:
correlation analysis of Tumor marker and therapeutic effect | 3 years
  Tumor markers include PD-L1、TMB、MSI、dMMR

CONTACTS AND LOCATIONS:
Locations (1):
- Shaohong Yin, Linyi, Shandong, China